CLINICAL TRIAL: NCT01077193
Title: Surgical Intervention in Bariatric Patients: Excess Weight Loss in the Morbidly Obese Following Gastric Plication
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to commercial considerations and potential patient attrition at 3 years. There were no patient safety or procedure efficacy reasons.
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-09-0006
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Morbid Obesity
Keywords: Bariatric; Obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gastric Plication Surgery (Other)
  Interventions: Procedure: Gastric Plication

INTERVENTIONS:
Procedure: Gastric Plication — A laparoscope will be inserted to visualize the surgical area and confirm absence of injury to any surrounding organ or structure. A flexible endoscope will be passed transorally into the gastric lumen to provide insufflation.
  The greater curvature of the stomach is separated from the greater omentum using a harmonic scalpel starting approximately 3cm from the pylorus and ending at or near the angle of His. As needed, adhesions to the posterior surface of the stomach may be transected.
  At least two rows of at least five continuous stitches will be placed laparoscopically about the greater curvature of the stomach starting at or near the angle of His and ending in the antrum. An endoscope will be used to maintain a lumen during the procedure, ensuring one exists after the procedure.

SUMMARY:
Up to 45 men and women who meet the entry criteria will undergo the gastric plication procedure. The study will assess subject excess weight loss (%EWL) following the study procedure at 1, 3, 6, 12, 18, 24, 30 and 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing to give consent and comply with evaluation and treatment schedule (for female patients, this includes agreement to use a reliable (per investigator) form of birth control for the duration of the trial);
2. 18 to 65 years of age (inclusive);
3. Subject meets ASMBS and NIH criteria: (consensus.nih.gov)

   BMI ³ 40 kg/m2 and £ 50 kg/m2; or, BMI 35-40 kg/m2 with one or more significant co-morbid medical conditions which are generally expected to be improved, reversed, or resolved by weight loss, including:
   * Hyperlipidemia
   * Mild obstructive sleep apnea (per Investigator discretion)
   * Hypertension
   * Osteoarthritis of the hip or knee per investigational site's criteria for which the subject is being treated;
4. ASA Class I - III;
5. Agree to refrain from any type of weight-loss drug (prescription or OTC) or elective procedure that would affect body weight for the duration of the trial;
6. HbA1C < 11%; and
7. For subjects who have Type 2 diabetes, medication regimen is no more complex (2 oral medications) than oral metformin plus one oral sulfonylurea plus once daily insulin injection.

Exclusion Criteria:

1. Documented history of drug and/or alcohol abuse within two (2) years of the Screening Visit;
2. Previous malabsorptive or restrictive procedures performed for the treatment of obesity;
3. Scheduled concurrent surgical procedure, with the exception of SOC liver biopsy;
4. Women of childbearing potential who are pregnant or lactating at the time of screening or at the time of surgery;
5. Psychiatric disorders that may affect compliance with the clinical trial, including dementia, active psychosis, severe depression requiring > 2 medications, or history of suicide attempts;
6. Participation in any other investigational device or drug study (non-survey based trial; long-term enrollment in such studies as requiring periodic laboratory tests, etc., would be allowed) within 12 weeks of enrollment;
7. Any condition which precludes compliance with the study, including:

   1. Inflammatory diseases of the gastrointestinal tract, including severe intractable esophagitis, gastric ulceration, duodenal ulceration, or specific inflammation such as Crohn's disease or ulcerative colitis that have been active within the past 10 years;
   2. Congenital or acquired anomalies of the GI tract, including atresias or stenosis;
   3. Severe cardiopulmonary disease or other serious organic disease that makes the subject a high-risk surgical candidate;
   4. Uncontrolled hypertension;
   5. Portal hypertension;
   6. Chronic or acute upper gastrointestinal bleeding conditions (e.g., gastric or esophageal varices);
   7. Cirrhosis;
   8. Congenital or acquired intestinal telangiectasia;
   9. Esophageal or gastric disorders including moderate severe preoperative reflux, dysmotility, or Barrett's esophagus;
   10. Presence of hiatal hernia greater than 2cm in length, with the exception of a small sliding hiatal hernia previously undiagnosed and discovered during the surgical procedure;
   11. Prior surgery of the foregut including hiatal hernia repair or prior gastric surgery;
   12. Known history of clotting disorders, hemoglobinopathies, and hemolytic disorders, including pulmonary embolus and Deep Vein Thrombosis;
   13. Pancreatitis;
   14. Gallstones (confirmed via ultrasound);
   15. Immunocompromised such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders;
   16. Use of thiazolidinediones ("glitazones"), or
   17. Conditions that, in the opinion of the investigator, may jeopardize the subject's well-being and/or the soundness of this clinical study;
8. History or presence of pre-existing autoimmune connective tissue disease; and
9. Use of prescription or over the counter weight reduction medications or supplements within thirty days of the Screening Visit or the duration of study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
- OB Klinika, a.s., Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period began in October 2009 and ended in November 2010 at three sites (1 academic site, 2 medical clinics).
Pre-assignment Details: No significant events were involved - subjects were evaluated for inclusion and exclusion criteria and proceeded to surgery if they qualified. This is a 1-arm trial.
Groups:
- Gastric Plication Surgery: Gastric Plication : A laparoscope will be inserted to visualize the surgical area and confirm absence of injury to any surrounding organ or structure. A flexible endoscope will be passed transorally into the gastric lumen to provide insufflation.
  The greater curvature of the stomach is separated from the greater omentum using a harmonic scalpel starting approximately 3cm from the pylorus and ending at or near the angle of His. As needed, adhesions to the posterior surface of the stomach may be transected.
  At least two rows of at least five continuous stitches will be placed laparoscopically about the greater curvature of the stomach starting at or near the angle of His and ending in the antrum. An endoscope will be used to maintain a lumen during the procedure, ensuring one exists after the procedure.
Period: Overall Study
Arm/Group | Gastric Plication Surgery
Started | 44
Completed | 0
Not Completed | 44
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 1
Not completed — Study Terminated by Sponsor | 40

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population: All subjects who underwent the gastric plication surgery.
Arm/Group | Gastric Plication Surgery
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 29
  Czech Republic | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Excess Weight Loss at 3 Years With Last Observation Carried Forward
Description: Percent excess weight change from baseline to 3 years was calculated as (the baseline weight minus the weight at 3 years) divided by the (baseline weight minus the ideal body weight (using the upper limit of the midpoint range in the Metropolitan Tables for Life Insurance, 1983) x 100). Last observation carried forward was used for early terminated subjects.
  One-sided, alpha=0.025, t-test of the Percent Excess Weight Loss (EWL) at 3-years to demonstrate non-inferiority to the target weight loss value of 41.1%EWL
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: percentage of baseline excess weight
Arm/Group | Gastric Plication Surgery
Number analyzed (Participants) | 44
percentage of baseline excess weight | 37.9 (25.18)
Statistical Analysis 1: Comparison: Gastric Plication Surgery; A sample size of 32 achieves power>90% to demonstrate non-inferiority using a one-sided t-test (alpha=0.025) when the margin of equivalence is a 5% difference in EWL. The true difference between %EWL for patients undergoing a greater curvature procedure and the target %EWL is hypothesized to be 0. The target %EWL at 3 years is 41.1%, based upon prior studies. This power analysis assumes data are drawn from a single population with a standard deviation of 8.20; Test type: Non-Inferiority or Equivalence — See above; p = 0.3227, t-test, 1 sided — No multiple comparison adjustments are necessary as this is a single hypothesis on 1 parameter for a within group change comparison to 36.1%; Mean Percent Excess Weight Loss = 37.9, 95% CI 2-sided [30.2 to 45.5], Standard Deviation 25.18

ADVERSE EVENTS:
Arm/Group | Gastric Plication Surgery
Serious Adverse Events (participants affected / at risk) | 8/44
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Plication Surgery (N=44)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Gastric perforatin (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3)
Abdominal sepsis (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (3)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Plication Surgery (N=44)
Nausea (Gastrointestinal disorders) | 40 (45)
Abdominal pain (Gastrointestinal disorders) | 20 (25)
Procedural pain (Injury, poisoning and procedural complications) | 20 (20)
Vomiting (Gastrointestinal disorders) | 17 (19)
Body temperature increased (Investigations) | 8 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 4 (5)
Urinary tract infection (Infections and infestations) | 4 (4)
Hiatus hernia (Gastrointestinal disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (6)
Headache (Nervous system disorders) | 3 (7)
Hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed that the first publication should be made in conjunction with the presentation of a joint, multicenter publication with the PIs from all sites contributing data, analyses, and comments. If this publication was not submitted within 12 months after conclusion of the Study at all sites, termination of the Study at all sites, or after Sponsor confirmed there would be no multicenter Study publication, whichever is first, the PIs could publish the results from their individual sites.